CLINICAL TRIAL: NCT06668064
Title: A 2-year Phase 3, Multicenter, Prospective, Randomized, Double-Masked, Parallel-Group Study of EYP-1901, a Tyrosine Kinase Inhibitor (TKI), Compared to Aflibercept in Subjects With Wet AMD
Brief Title: A 2-year Study of EYP-1901 in Subjects With Wet Age Related Macular Degeneration (wAMD) (LUGANO) Primary Efficacy Will be Determined at Week 56
Acronym: wAMD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYP-1901-301
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Wet Age Related Macular Degeneration; wAMD
Keywords: Wet Age-related Macular Degeneration; Tyrosine Kinase Inhibitor; EYP-1901; EyePoint
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EYP-1901 2686 µg (Experimental): EYP-1901
  Interventions: Drug: EYP-1901
- Aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept (2.0 mg)

INTERVENTIONS:
Drug: EYP-1901 — Intravitreal Injection
  Arms: EYP-1901 2686 µg
Drug: Aflibercept (2.0 mg) — Intravitreal Injection
  Arms: Aflibercept

SUMMARY:
This is a phase 3 randomized, double -masked study comparing the efficacy of EYP-1901 against Aflibercept.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated or treatment naïve patients with a documented diagnosis of wAMD in the study eye, with onset of disease that began at any time prior to the Screening Visit.
* Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) letter score between 78 to 35 letters (approximately 20/32 to 20/200 Snellen equivalent) in the study eye at the Screening Visit and on Baseline (Day 1).
* For previously-treated subjects, must have been treated with at least 2 anti-VEGF IVT injections (i.e., aflibercept 2 mg, aflibercept 8 mg, bevacizumab, ranibizumab, or faricimab) in the previous 6 months for wAMD per standard of care in the study eye prior to the Screening Visit.

Exclusion Criteria:

* Subfoveal fibrosis, atrophy, or scarring in the center subfield.
* BCVA using ETDRS charts <20 letters (20/400 Snellen equivalent) in the fellow eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Average change in best corrected visual acuity (BCVA) | Weeks 52 and 56

SECONDARY OUTCOMES:
Rate of injection burden | Week 56
Average change in best corrected visual acuity (BCVA) | Week 96

CONTACTS AND LOCATIONS:
Locations (81):
- United States (81):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Partners of Northwest Arkansas, Springdale, Arkansas
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Macula and Retina Institute, Glendale, California
  - Retina Consultants San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - Bay Area Retina Associates, Walnut Creek, California
  - American Institute of Research, Whittier, California
  - RSC Research, PLLC, Denver, Colorado
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Advanced Vision Institute, Longmont, Colorado
  - Connecticut Eye Consultants, P.C., Danbury, Connecticut
  - SightSera Clinical Research LLC, Greenwich, Connecticut
  - Retina Group of New England, PC, Waterford, Connecticut
  - Advanced Research, LLC, Deerfield Beach, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Group of Florida, Sarasota, Florida
  - MedEye Associates, South Miami, Florida
  - Retina Specialists of Tampa, Tampa, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Gerogia Retina, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Retina Associates, Elmhurst, Illinois
  - University Retina and Macula Associates, Lemont, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Retina Associates LLC, Lenexa, Kansas
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Retina Groups of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Specialists, Towson, Maryland
  - Ophthalmic Consultants of Boston OCB - Boston, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Deep Blue Retina Clinical Research PLLC, Southaven, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - NJ Retina, Teaneck, New Jersey
  - NJ Retina, Toms River, New Jersey
  - Vision Research Center at Eye Associates of New Mexico, Albuquerque, New Mexico
  - Retina Vitreous Surgeons of CNY, PC, Liverpool, New York
  - Retina Associates of Western NY, PC, Rochester, New York
  - Retina Consultants PLLC, Slingerlands, New York
  - Western Carolina Retinal Associates, PA, Asheville, North Carolina
  - Cape Fear Retinal Associates, PC, Wilmington, North Carolina
  - Piedmont Retina Specialists, P.A. - Winston-Salem Office, Winston-Salem, North Carolina
  - Midwest Retina, Inc., Dublin, Ohio
  - Tulsa Retina Consultant, Tulsa, Oklahoma
  - Verum Research LLC, Eugene, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Eye Care Specialists - Kingston Location, Kingston, Pennsylvania
  - Retina Consultants, Charleston, South Carolina
  - Palmetto Retina Center, Florence, South Carolina
  - Retina Consultants of Carolina P.A, Greenville, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Research Institute of Texas Integrated Clinical Research, Abilene, Texas
  - Retina and Vitreous of Texas, Bellaire, Texas
  - Retina Consultants of Texas (Retina Consultants of Houston) - Woodlands, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Houston Eye Associates, Houston, Texas
  - Texas Retina Associates, Plano, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Retinal Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Tyler Retina Consultants, Tyler, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Salt Lake Retina, West Jordan, Utah
  - The Retina Group of Washington, Fairfax, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Retina Associates, P.C., Winchester, Virginia
  - University of Wisconsin School of Medicine and Public Health (UWSMPH), Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided